CLINICAL TRIAL: NCT03428971
Title: P-wave Terminal Force in Patients With Atrial Fibrillation: Can we Predict Number of Hospitalisations and Left Atrial Electrical Remodelling? - Ptf-AF Trial
Brief Title: P-wave Terminal Force in Patients With Atrial Fibrillation.
Acronym: Ptf-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Maciej Wójcik, MD, PhD, Assistant Professor, Medical University of Lublin
Other Study IDs: MW-MULublin-1
Record Dates: First submitted 2018-02-02; First posted 2018-02-12 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; p-wave; hospitalization
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardioversion — Direct current (DC) cardioversion for sinus rhythm restoration

SUMMARY:
It is suggested that P-wave terminal force (Ptf), a product of the amplitude (PAM) and the duration (PT) of the terminal phase of P-wave in lead V1, shows early delay in left atrial conduction, observed earlier that the dilatation of left atrium.

The aim is to follow PT, PAM and Ptf changes during 5-year follow-up (5FU) and examine the relation of these changes to the number of AF episodes requiring hospitalisation (HOSP) for restoration of sinus rhythm (RSR).

DETAILED DESCRIPTION:
Background. It is suggested that P-wave terminal force (Ptf), a product of the amplitude (PAM) and the duration (PT) of the terminal phase of P-wave in lead V1, shows early delay in left atrial conduction, observed earlier that the dilatation of left atrium.

Aim. We aim to follow PT, PAM and Ptf changes during 5-year follow-up (5FU) and examine the relation of these changes to the number of AF episodes requiring hospitalisation (HOSP) for restoration of sinus rhythm (RSR).

We hypothesise that, in patients with atrial fibrillation (AF):

1. the index parameters (PT, PAM, Ptf), characterising left atrial repolarization, correlates the number of future hospitalisations (HOSP) aimed for restoration of sinus rhythm (RSR) in 5-year follow-up (5FU)
2. in 5FU the number of HOSP aimed for RSR correlates with the progression of left atrium electrical remodelling, expressed as PAM5,PT5, Ptf5 at 5FU.

ELIGIBILITY:
Inclusion Criteria:

* documented atrial fibrillation at admission
* successful restoration of sinus rhythms documented in 12-leads ECG,
* follow-up => 5 years

Exclusion Criteria:

* arrhythmia other than atrial fibrillation at admission,
* unsuccessful restoration of sinus rhythms,
* successful restoration of sinus rhythms but missing 12-leads ECG recording,
* previous ablation/operation within left atrium,
* follow-up < 5 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation admitted between 1.1.2001 and 30.12.2012 for elective and emergency hospitalization aimed for restoration of sinus rhythms with DC cardioversion.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-07 (Estimated); Study Completion 2020-12-07 (Estimated)

PRIMARY OUTCOMES:
Changes of P-wave time (PT), P-wave amplitude (PAM) and Ptf (P wave terminal force terminal V1-lead ) in 5-year follow-up (5FU). | 5 years
  All measurements based on ECG recording during sinus rhythm only.
  * "P-wave time (PT)" defined as time (measured in milliseconds, [ms]) of negative deflection of P wave in V1 lead of the standard 12-lead ECG;
  * "P-wave amplitude (PAM)" defined as maximum amplitude (measured in millivolts, [mV]) of negative deflection of P wave in V1 lead of the standard 12-lead ECG;
  * "P-wave terminal force (Ptf)" is a product of the amplitude and the duration of the terminal phase of P-wave in lead V1; Ptf = PT x PAM [ms x mV];
  * PT and PAM measured at index is defined as PT0 and PAM0, respectively
  * Calculated Ptf as a product of PT0 and PAM0 is defined as Ptf0;
  * PT and PAM measured at 5FU is defined as PT5 and PAM5, respectively;
  * Calculated Ptf as a product of PT5 and PAM5 is defined as Ptf5;
  * The change between PT0 and PT5 (PTC = PT5 - PT0) , PAM0 and PAM5 (PAMC = PAM5 - PAM0), Ptf0 and Ptf5 (PtfC = Ptf5 - Ptf0) will be calculated for each patient;

SECONDARY OUTCOMES:
Correlation between index PT0, PAM0, Ptf0 and number of hospitalizations (HOSP) in 5-year follow-up | 5 years
  Statistical analysis of Correlation between index PT0, PAM0, Ptf0 and number of hospitalizations (HOSP) in 5-year follow-up
Correlation between number of hospitalizations (HOSP) in 5- year follow-up and final PT5, PAM5, Ptf5 at the end of 5-year follow-up period. | 5 years
  Statistical analysis of Correlation between number of hospitalizations (HOSP) in 5- year follow-up and final PT5, PAM5, Ptf5 at the end of 5-year follow-up period.
Correlation between changes of PT, PAM, Ptf (PTC, PAMC, PtfC) and number of hospitalizations (HOSP) in 5-year follow-up. | 5 years
  Statistical analysis of Correlation between changes of PTC, PAMC, PtfC and number of hospitalizations (HOSP) in 5-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Wójcik, MD, PhD, Principal Investigator — Medical University of Lublin, Poland
Locations (1):
- Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wojcik M, Kuniss M, Berkowitsch A, Neumann T. P-wave terminal force and atrial fibrillation: a lesson learned from old masters. Rev Esp Cardiol (Engl Ed). 2012 Jun;65(6):584-5; author reply 585. doi: 10.1016/j.recesp.2012.01.015. Epub 2012 Mar 31. No abstract available. PMID 22465604
- [Background] Janin S, Wojcik M, Kuniss M, Berkowitsch A, Erkapic D, Zaltsberg S, Ecarnot F, Hamm CW, Pitschner HF, Neumann T. Pulmonary vein antrum isolation and terminal part of the P wave. Pacing Clin Electrophysiol. 2010 Jul;33(7):784-9. doi: 10.1111/j.1540-8159.2010.02754.x. Epub 2010 Mar 29. PMID 20374516
- [Background] Ishida K, Hayashi H, Miyamoto A, Sugimoto Y, Ito M, Murakami Y, Horie M. P wave and the development of atrial fibrillation. Heart Rhythm. 2010 Mar;7(3):289-94. doi: 10.1016/j.hrthm.2009.11.012. Epub 2009 Nov 12. PMID 20133209
- [Background] Martin Garcia A, Jimenez-Candil J, Hernandez J, Martin Garcia A, Martin Herrero F, Martin Luengo C. P wave morphology and recurrence after cardioversion of lone atrial fibrillation. Rev Esp Cardiol (Engl Ed). 2012 Mar;65(3):289-90. doi: 10.1016/j.recesp.2011.04.023. Epub 2011 Jul 30. No abstract available. English, Spanish. PMID 21803476